CLINICAL TRIAL: NCT01720147
Title: Quercetin in Children With Fanconi Anemia; a Pilot Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2011-2049; 1R01FD004383-01A1 (FDA)
Record Dates: First submitted 2012-07-25; First posted 2012-11-02 (Estimated); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Fanconi Anemia
Keywords: Fanconi Anemia; FA; Quercetin
MeSH Terms: conditions — Fanconi Anemia | interventions — Quercetin; Dietary Supplements

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Quercetin - Dietary Supplement (Experimental): Quercetin will be given orally on a twice a day schedule starting with weight adjusted dose for a maximum total daily dose of 1500 mg/day, for 4 months (16 weeks). Pharmacokinetics (PK) data will be analyzed after each cohort of 3 patients and will be used to optimize the dosing schedule (if required) for subsequent patients.
  An expansion cohort has been added to the study protocol. Up to 20 patients may be enrolled. The dose utilized will be the same as the max weight adjusted dose that showed biological activity in our last cohort of patients (subjects #10-12 from above).
  Interventions: Drug: Quercetin (dietary supplement)

INTERVENTIONS:
Drug: Quercetin (dietary supplement) — Quercetin will be given orally on a twice a day schedule starting with weight adjusted dose for a maximum total daily dose of 1500 mg/day, for 4 months (16 weeks). Pharmacokinetics (PK) data will be analyzed after each cohort of 3 patients and will be used to optimize the dosing schedule (if required)for subsequent patients.
  An expansion cohort has been added to the study protocol. Up to 20 patients may be enrolled. The dose utilized will be the same as the max weight adjusted dose that showed biological activity in our last cohort of patients (subjects #10-12 from above).

SUMMARY:
Fanconi anemia (FA) is an autosomal recessive disease characterized by progressive bone marrow failure (BMF), congenital abnormalities and a predisposition to malignancy.

DETAILED DESCRIPTION:
Current therapies for children with Fanconi anemia (FA) and bone marrow failure, i.e. androgens or bone marrow transplantation, are associated with significant morbidity and mortality.

This is a pilot study aiming to assess feasibility, toxicity and pharmacokinetics of oral Quercetin therapy in patients with FA. This is a first step towards a clinical study of the efficacy of Quercetin therapy in delaying progression of BMF in FA.

Additional correlative studies will include assessment of impact of Quercetin on reduction of Reactive Oxygen Species (ROS), maintenance or improvement of hematopoietic stem cell (HSC) reserve, improvement of hematopoiesis (i.e. peripheral counts) and insulin sensitivity/glucose tolerance.

This study is an open-label single arm study.

Funding Source - FDA OOPD

Accrual closed for the main study. Expansion cohort added to observe additional patients at the desired dose.

Expansion Cohort:

The second and third cohort of participants completed the study treatment as expected, tolerating Quercetin well without any DLT. Based on the PK and ROS analyses, the dose was increased for the fourth cohort (subjects #10-12). To observe additional patients at the desired dose, an expansion cohort is being added. Up to 20 patients will be enrolled in the expansion cohort. The purpose of the expansion cohort is to assess the effects of quercetin supplement at the desired dose on clinical and biological endpoints.

Patients in the expansion cohort will receive quercetin treatment for the first 26 weeks. Patients will be able to continue quercetin supplement after the completion of the study period of 26 weeks if they wish. If patients decide to continue quercetin after the first 26 weeks, quercetin will be provided by the investigational pharmacy for up to 1 year. Patients who continue quercetin supplement after 26 weeks, but discontinue quercetin before 1 year will be followed through the 1 year visit. Patients who discontinue quercetin supplement any time after the 1 year visit will be followed through the 2 year visit.

Patients previously enrolled in the initial phase of the study (cohorts 1-4) may be considered for enrollment on the expansion cohort of the study provided they meet all inclusion and exclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of FA proven by DEB test or molecular testing
* Able to take enteral medication
* All age groups, including adults

Exclusion Criteria:

* Patients with morphological evidence of myelodysplasia or leukemia
* Renal failure requiring dialysis
* Total bilirubin > 3 mg/dl and/or SGPT >200 at time of enrollment
* Patients who are pregnant or breastfeeding or are at risk of pregnancy and are unable to use acceptable methods of birth control during the length of the study
* Patients receiving cyclosporine or digoxin therapy or are unable to discontinue either treatment due to medical reasons
* Patients who have received quercetin supplementation or other antioxidants within the last 30 days

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-07; Primary Completion 2021-10-26 (Actual); Study Completion 2021-10-26 (Actual)

PRIMARY OUTCOMES:
Measure the ability to administer twice daily oral quercetin therapy in patients with Fanconi Anemia (FA). | 4 months (16 weeks)
Measure safety of oral quercetin therapy in patients with FA | 4 months (16 weeks)
To measure pharmacokinetics (PK) of oral quercetin therapy in patients with FA | 4 months (16 weeks)

SECONDARY OUTCOMES:
To measure the impact of quercetin therapy on reduction of Reactive Oxygen Species (ROS). | 4 months (16 weeks) and 1 year
Number of participants with improved hematopoiesis. | 4 months (16 weeks) and 1 year
Measure the preservation of hematopoietic stem cell reserve in patients with FA | 4 months (16 weeks) and 1 year
To measure the impact of quercetin therapy on changes in insulin sensitivity/glucose tolerance. | 4 month (16 weeks) and 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Parinda Mehta, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mehta PA, Nelson A, Loveless S, Lane A, Fukuda T, Teusink-Cross A, Elder D, Lagory D, Miller E, Cancelas JA, Howell J, Zhao J, Mizuno K, Myers KC, Lake K, McIntosh K, Setchell KDR, Luebbering N, Edwards S, Chihanga T, Wells SI, Davies SM. Phase 1 study of quercetin, a natural antioxidant for children and young adults with Fanconi anemia. Blood Adv. 2025 Apr 22;9(8):1927-1939. doi: 10.1182/bloodadvances.2024015053. PMID 39820512